CLINICAL TRIAL: NCT01227720
Title: Comparative Pharmacokinetic Study of New Oral Nicotine Replacement Therapy Products - A Study in Healthy Smokers.
Brief Title: Comparative Pharmacokinetic Study of New Oral Nicotine Replacement Therapy Products.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McNeil AB (Industry)
Responsible Party: Sponsor
Organization: Johnson & Johnson Consumer and Personal Products Worldwide (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NICTDP1076
Record Dates: First submitted 2010-10-22; First posted 2010-10-25 (Estimated); Last update posted 2012-07-10 (Estimated); Status verified 2012-07

CONDITIONS: Tobacco Dependence
Keywords: Smoking Cessation, Nicotine pharmacokinetics
MeSH Terms: conditions — Tobacco Use Disorder; Smoking Cessation | interventions — Nicotine Replacement Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- A NSL2L (Experimental): Experimental Nicotine Replacement Therapy (NRT)(L) 2 mg
  Interventions: Drug: Experimental Nicotine Replacement Therapy (NRT) 2 mg
- B Lozenge (Active Comparator): Marketed Nicotine Lozenge 2 mg
  Interventions: Drug: Marketed Nicotine Lozenge
- C NSL4M (Experimental): Experimental NRT (M) 4 mg
  Interventions: Drug: Experimental Nicotine Replacement Therapy (NRT)
- D Lozenge (Active Comparator): Marketed Nicotine Lozenge 4 mg
  Interventions: Drug: Marketed Nicotine Lozenge
- E NSL4L (Experimental): Experimental NRT (L) 4 mg
  Interventions: Drug: Experimental Nicotine Replacement Therapy (NRT)
- F NSL4H (Experimental): Experimental NRT (H) 4 mg
  Interventions: Drug: Experimental Nicotine Replacement Therapy (NRT)

INTERVENTIONS:
Drug: Experimental Nicotine Replacement Therapy (NRT) 2 mg — 2 mg Single-dose of new NRT product (NSL2L)
  Other Names: Not yet marketed
  Arms: A NSL2L
Drug: Experimental Nicotine Replacement Therapy (NRT) — 4 mg Single-dose of new NRT product
  Other Names: Not yet marketed
  Arms: C NSL4M; E NSL4L; F NSL4H
Drug: Marketed Nicotine Lozenge — 2 mg Single-dose of marketed lozenge
  Other Names: NiQuitin™ lozenge
  Arms: B Lozenge
Drug: Marketed Nicotine Lozenge — 4 mg Single-dose of marketed lozenge
  Other Names: NiQuitin™ lozenge
  Arms: D Lozenge

SUMMARY:
Comparative pharmacokinetic study of new oral nicotine replacement therapy products.

DETAILED DESCRIPTION:
This study compares new oral Nicotine Replacement Therapy (NRT) products containing 2 and 4 mg nicotine with NiQuitin™ lozenge 2 mg and 4 mg, after 12 hours of nicotine abstinence, with respect to nicotine pharmacokinetics, during 12 hours after start of administration. Single doses of treatment A, B, C, and D are given once in the morning during separate treatment visits scheduled in a crossover setting with randomized treatment sequences, also including a fifth treatment visit with either treatment E or F. The study will include 104 healthy smokers between the ages of 19 and 50 years, who have been smoking at least 10 cigarettes daily during at least one year preceding inclusion. The study will be performed at two sites with 52 subjects at each site. Subjects and study personnel will be aware of which treatment is administered at a given visit.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects, smoking at least 10 cigarettes daily during at least one year preceding inclusion and BMI between 17.5 and 30.0 kg/m2.
* Female participants of child-bearing potential are required to use a medically acceptable means of birth control.
* A personally signed and dated informed consent document, indicating that the subject has been informed of all pertinent aspects of the study.

Exclusion Criteria:

* Pregnancy, lactation or intended pregnancy.
* Treatment with an investigational product or donation or loss of blood within 3 month preceding the first dose of study medication.

Ages: 19 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 104 (Actual)
Dates: Start 2009-08; Primary Completion 2009-12 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Maximum Plasma Concentration | during 12 hours after product administration
  The maximum observed nicotine concentration in plasma (Cmax)
Area under the Curve | after 12 hours
  The area under the plasma concentration-vs-time curve until the last measurable concentration (AUCt) and the area under the plasma concentration-vs.-time curve until infinity (AUC∞)

SECONDARY OUTCOMES:
Time of Maximum Concentration | during 12 hours after start of product administration
  The time of occurrence of maximum concentration (Tmax)
Terminal Elimination Rate Constant | during 12 hours after start of product administration
  The terminal nicotine elimination rate constant (λz)
Oral Dissolution Time | from administration until completely dissolved
  Actual time required for oral dissolution

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth Kruse, PhD, Study Director — McNeil AB
Locations (2):
- Sweden (2):
  - Lund University Hospital Clinical Trial Unit, Lund
  - McNeil AB Clinical Pharmacology R&D, Lund